CLINICAL TRIAL: NCT07403942
Title: Cosmetic Efficacy Testing
Brief Title: The Skin Anti-Aging Effects of Vitamin K2 (MK-7): a Clinical Split-Face/Neck Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Ascend Biotech Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2024-293-ZH-262
Record Dates: First submitted 2026-01-29; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Skin Aging of Face and Neck
Keywords: Vitamin K2; MK-7; Skin Aging
MeSH Terms: interventions — Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Face-and-Neck Cream (Placebo Comparator): Participants apply the Placebo Face-and-Neck Cream (base formulation without Vitamin K2) to the contralateral half of the face and neck. Used twice daily (morning and evening) for 8 weeks.
  Interventions: Other: Placebo Face-and-Neck Cream
- Face-and-Neck Cream (Active Comparator): Participants apply the Face-and-Neck Cream (containing 0.05% Vitamin K2) to one randomly assigned half of the face and neck. Used twice daily (morning and evening) for 8 weeks.
  Interventions: Other: Face-and-Neck Cream (with 0.05% Vitamin K2)

INTERVENTIONS:
Other: Face-and-Neck Cream (with 0.05% Vitamin K2) — This is a topical cosmetic cream (face and neck cream) containing 0.05% BioYoung™ MK-7 (Vitamin K2) as the key active ingredient. The product is a white to light yellow cream, supplied in plastic bottles. Each participant applies this cream to one randomly assigned half of the face and neck. The application regimen is twice daily (morning and evening), using approximately 0.5g per application, for a duration of 8 weeks.
  Other Names: Face-and-Neck Cream (with 0.05% BioYoung™ MK-7)
  Arms: Face-and-Neck Cream
Other: Placebo Face-and-Neck Cream — This is the control topical cosmetic cream (face and neck cream). It is the base formulation identical to the test cream but without the addition of Vitamin K2. The product is a white to light yellow cream, supplied in plastic bottles. Each participant applies this cream to the contralateral half of the face and neck (opposite to the test product side). The application regimen is twice daily (morning and evening), using approximately 0.5g per application, for a duration of 8 weeks.
  Arms: Placebo Face-and-Neck Cream

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of a facial and neck cream containing Vitamin K2 in improving skin hydration, elasticity, firmness, and reducing wrinkles in 36 female participants aged 35-60 years with concerns of facial dryness, dullness, laxity, and neck lines. The main questions it aims to answer are:

Does the test cream significantly improve skin hydration (Corneometer), reduce transepidermal water loss (Vapometer), and enhance skin elasticity and firmness (Cutometer) compared to a control cream?

Does the test cream significantly reduce wrinkle severity (assessed by Rz and Ra parameters via AEVA-HE rapid optical imaging) in areas including the neck, cheeks, marionette lines, and crow's feet compared to a control cream?

Researchers will compare the test cream (applied to one randomized half-face and neck) to the control cream (applied to the contralateral half-face and neck) to see if the test cream demonstrates superior efficacy in improving the measured skin parameters.

Participants will:

Apply the test cream to one assigned side of the face and neck, and the control cream to the other side, twice daily for 8 weeks.

Attend evaluation visits at baseline, 2, 4, and 8 weeks for instrumental measurements (skin hydration, TEWL, elasticity, rapid optical imaging, facial imaging) and to complete subjective questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Is a Chinese female aged between 35 and 60 years (inclusive).
* Presents with facial skin concerns including dryness, dullness, and laxity.
* Has crow's feet (outer canthus wrinkles) with a visual assessment grade of 2 to 4 (on a 0-6 scale).
* Self-reports concerns about neck wrinkles.
* Is in good general health at the time of screening.
* Is willing and able to provide written informed consent.
* Is willing and able to comply with all study procedures and product usage requirements for the duration of the study.

Exclusion Criteria:

* Is planning pregnancy, is pregnant, lactating, or within 6 months postpartum.
* Has a history of severe systemic diseases, immunodeficiency, or autoimmune diseases.
* Has a history of allergic diseases or has experienced cosmetic allergies within the past 1-2 years.
* Has had dermatological diseases on the test areas (face and neck) or is undergoing related medical treatment within the past 3 months.
* Has an active cold, influenza, or other acute illness at the study start that may affect participation.
* Is currently participating, or has participated within the past month, in another clinical study involving the test areas.
* Is deemed unsuitable for participation by a dermatologist's assessment.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-12-26 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Change in Facial Skin Elasticity (R0, R1 and F4) | At Baseline, Week 2, Week 4, and Week 8
  Assessed using a Cutometer MPA580.Measurements are taken on the cheek area. R0 (Uf) represents the maximum skin deformation under suction. A lower R0 value indicates greater resistance to tensile deformation, reflecting superior skin firmness.
  R1 (Uf - Ua) quantifies the immediate elastic recovery after suction release. A lower R1 value signifies faster restoration to baseline morphology, demonstrating enhanced skin elasticity.
  F4, the viscoelastic fatigue parameter, quantifies energy dissipation during cyclic skin deformation. A lower F4 value indicates enhanced viscoelastic integrity of the skin.
Change in Roughness Parameters (Ra and Rz ) of Face and Neck Wrinkles | At Baseline, Week 2, Week 4, and Week 8
  Assessed by AEVA-HE rapid optical imaging system. Ra represents the arithmetic average of absolute deviations of skin surface profile points from the mean line across the entire assessment length. It quantifies the overall smoothness of the skin surface. Lower Ra values indicate smoother skin with less pronounced wrinkle formation.
  Rz is calculated by dividing the skin surface profile into five equal sampling lengths. The parameter represents the arithmetic mean of the distances between the highest peaks and deepest valleys within each segment, quantifying the extreme variations in skin surface topography. As a key indicator of macro-textural irregularities, lower Rz values correspond to reduced skin unevenness.
Change in Facial Sagging (Mandibular Plane Angle) | At Baseline, Week 2, Week 4, Week 8
  Quantified by analyzing standard white-light photographs taken with a VISIA imaging system. The mandibular plane angle is measured in degrees (°) using image analysis software (Image-Pro Plus). An increase in the angle indicates a sharper, more defined, and firmer jawline contour.

SECONDARY OUTCOMES:
Change in Skin Hydration | At Baseline, Week 2, Week 4, Week 8
  Measured by a Corneometer CM825 on the cheek. Values are expressed in arbitrary units (a.u.). A higher value indicates better skin hydration.
Change in Facial Transepidermal Water Loss (TEWL) | At Baseline, Week 2, Week 4, Week 8
  Measured in grams per square meter per hour (g/m²h) using a standardized vapometer (Vapometer, SWL5201) under controlled environmental conditions (21 ± 1°C, 50 ± 10% RH). Measurements were taken on the cheek area (zygomatic region). A lower value indicates reduced water loss and improved skin barrier function.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Sino-German Union Cosmetic Institute Co., Ltd., Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF